CLINICAL TRIAL: NCT02701114
Title: A Comparison of Proximal Versus Distal Continuous Adductor Canal Blocks After Total Knee Arthroplasty
Brief Title: Proximal Versus Distal Adductor Canal Blocks for Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Principal Investigator, Neil Hanson, Staff Anesthesiologist, Benaroya Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB15118
Record Dates: First submitted 2016-02-29; First posted 2016-03-08 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proximal (Active Comparator): Proximal Adductor Canal Block
  Interventions: Procedure: Proximal Adductor Canal Block
- Distal (Active Comparator): Distal Adductor Canal Block
  Interventions: Procedure: Distal Adductor Canal Block

INTERVENTIONS:
Procedure: Proximal Adductor Canal Block — Continuous Nerve Block
  Arms: Proximal
Procedure: Distal Adductor Canal Block — Continuous Nerve Block
  Arms: Distal

SUMMARY:
This study is designed to evaluate pain control of continuous adductor canal blocks placed proximally versus distally within the canal. The investigators hypothesize that there will be similar pain control between both groups.

DETAILED DESCRIPTION:
This study is a non-inferiority trial designed to determine whether placement of a continuous block within the adductor canal has a substantial impact on pain following total knee arthroplasty. Our primary outcome to determine this difference will be opioid consumption within the first day following surgery. Secondary outcomes will include: pain scores, quadriceps strength, and distance ambulated during physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral Total Knee Arthroplasty
* ASA physical status I-III
* >18 years old
* Non-pregnant
* Consent to participate in the study

Exclusion Criteria:

* Refusal to participate
* <18 years old
* Chronic opioid use
* Localized infection Pregnancy Pre-existing coagulopathy Allergy to ultrasound gel or local anesthetics Contraindication to or refusal of spinal anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption (IV Morphine Equivalents) | 24 Hours
  Total opioid consumption

SECONDARY OUTCOMES:
Opioid Consumption (IV Morphine Equivalents) | 48 Hours
  Total opioid consumption
Pain (Numeric Rating) | 48 Hours
  NRS Pain Scale
Quadriceps Strength (% of Baseline) | 48 Hours
  Maximum Isometric Voluntary Contraction
Distance Ambulated (Feet) | 48 Hours
  Total distance ambulated during physical therapy

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Hanson, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Meier AW, Auyong DB, Yuan SC, Lin SE, Flaherty JM, Hanson NA. Comparison of Continuous Proximal Versus Distal Adductor Canal Blocks for Total Knee Arthroplasty: A Randomized, Double-Blind, Noninferiority Trial. Reg Anesth Pain Med. 2018 Jan;43(1):36-42. doi: 10.1097/AAP.0000000000000692. PMID 29140959